CLINICAL TRIAL: NCT02262845
Title: A Prospective Multi-Center Registry Using Plastic Pancreatic Stents for Short Term Drainage of the Pancreatic Duct
Brief Title: Short Term Pancreatic Stenting Registry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90987979
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Post-ERCP Acute Pancreatitis; Pancreatic Duct Stricture; Pancreatic Duct Stones; Pancreatic Duct Leakage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Group A: PEP Risk: In subjects deemed at high risk for acute pancreatitis post-endoscopic retrograde cholangiopancreatography (ERCP)
  Interventions: Device: The Advanix™ Pancreatic Stent and NaviFlex RX Pancreatic Delivery System and Pushers
- Group B: Impaired Pancreatic Duct Drainage: In subjects with a pancreatic duct stricture and/or pancreatic duct stones and/or pancreatic duct sludge or debris, possibly, but not exclusively before or after ESWL or before pancreatic surgery
  Interventions: Device: The Advanix™ Pancreatic Stent and NaviFlex RX Pancreatic Delivery System and Pushers
- Group C: Pancreatic Duct Leak: In subjects with a pancreatic duct leak
  Interventions: Device: The Advanix™ Pancreatic Stent and NaviFlex RX Pancreatic Delivery System and Pushers
- Group D: Post Pancreatic Surgery: In subjects at risk of pancreatic duct leak or strictures after resection of a pancreatic lesion close to the main pancreatic duct or at the level of the pancreatico-jejunostomy after pancreatico-duodenectomy
  Interventions: Device: The Advanix™ Pancreatic Stent and NaviFlex RX Pancreatic Delivery System and Pushers
- Group E: Other: In subjects with other indications
  Interventions: Device: The Advanix™ Pancreatic Stent and NaviFlex RX Pancreatic Delivery System and Pushers

INTERVENTIONS:
Device: The Advanix™ Pancreatic Stent and NaviFlex RX Pancreatic Delivery System and Pushers — Used to drain pancreatic ducts

SUMMARY:
The purpose of this study is to document clinical utility and distribution of indications for short term pancreatic stenting, and stent type preference by indication at tertiary referral centers with expertise in pancreatic endotherapy.

DETAILED DESCRIPTION:
The study is designed as an all-comer, prospective, multi-center, consecutive cohort series, open-label study.

Detailed objective: To confirm the clinical utility of Advanix™ Pancreatic Stents when used per standard of practice to facilitate pancreatic duct drainage in the following clinical presentations:

* Group A: PEP Risk - In subjects deemed at high risk for acute pancreatitis post-endoscopic retrograde cholangiopancreatography (ERCP)
* Group B: Impaired Pancreatic Duct Drainage - In subjects with a pancreatic duct stricture and/or pancreatic duct stones and/or pancreatic duct sludge or debris, possibly, but not exclusively before or after ESWL or before pancreatic surgery
* Group C: Pancreatic Duct Leak - In subjects with a pancreatic duct leak
* Group D: Post Pancreatic Surgery - In subjects at risk of pancreatic duct leak or strictures after resection of a pancreatic lesion close to the main pancreatic duct or at the level of the pancreatico-jejunostomy after pancreatico-duodenectomy
* Group E: Other - In subjects with other indications

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 18 or older.
2. Subjects who require pancreatic drainage and are amenable to endoscopic techniques.
3. Subjects willing and able to comply with the study procedures and follow up schedule and willing to provide written informed consent to participate in the study.
4. Subjects satisfying at least one of the following clinical presentations:

   1. high risk of acute pancreatitis post ERCP
   2. impaired pancreatic duct drainage and pain associated with a pancreatic duct dominant stricture and/or stones and/or sludge/debris, possibly before ESWL or before pancreatic surgery
   3. need to maintain proper pancreatic duct drainage in the presence of a pancreatic duct leak
   4. need to maintain proper pancreatic duct drainage after surgical resection of a pancreatic lesion close to the main pancreatic duct or at the level of the pancreatico-jejunostomy after pancreatico-duodenectomy

Exclusion Criteria:

1. Subjects for whom endoscopic techniques are contraindicated.
2. Subjects with known sensitivity to any components of the stents or delivery systems.
3. Subjects with coagulopathy outside of what is deemed acceptable for ERCPs per standard of practice
4. Subjects who are currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor.
5. Subjects unable or refusing to comply with the follow-up schedule including subject living at such a distance from the investigational center that attending follow-up visits would be unusually difficult or burdensome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will examine how well the Advanix Pancreatic stent helps drainage of the pancreas when used per standard-of-practice in many different situations.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Clinical Success: Group A (PEP Risk) | Stent placement through 48 hours post stent placement
  Absence of acute pancreatitis from stent placement through 48 hours post stent placement
Clinical Success: Group B (Impaired Pancreatic Duct Drainage) | Stent placement through stent removal
  Absence of acute pancreatitis from stent placement through stent removal and, where applicable, improvement of pain at stent removal compared to baseline
Clinical Success: Group C (Pancreatic Duct Leak): | Stent Removal
  Resolution of pancreatic duct leak at stent removal
Clinical Success: Group D (Post Pancreatic Surgery) | Stent Removal
  Absence of pancreatic duct leak and stricture at stent removal
Clinical Sucess: Group E (Other) | Stent Removal
  Resolution of the indication for stent placement at stent removal

SECONDARY OUTCOMES:
Serious Adverse Events and all occurrences of acute pancreatitis | Through end of study
  Occurrence and severity of serious adverse events related to the stent and/or the stent placement and/or stent removal procedures as applicable and all occurrences of acute pancreatitis.
Technical Success | Stent Placement
  Evaluation of technical success defined as the ability to place the stent in a satisfactory position in the main pancreatic duct as determined by fluoroscopy.
Ease of use | Stent Placement
  Evaluation of ease of use documenting overall ease of placement, pushability of stent and ability to visualize the stent fluoroscopically.
Removability | Stent Removal
  Evaluation of removability defined as ability to remove the Advanix stent endoscopically without serious stent removal related adverse events.
Stent Migration | Through end of study
  Documentation of stent migration rates overall, by Group, and by stent type
Reintervention | Through end of study
  Evaluation of the occurrence of reintervention defined as any type of endoscopic, percutaneous, or surgical procedure to aid drainage of the pancreas after initial stent placement through end of follow-up.
Stent type preference | Stent Placement
  Documenting stent type preference by subject presentation and pancreatic plastic stenting indication.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Tarnasky, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (7):
- United States (4):
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Methodist Dallas Medical Center, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Evangelisches Krankenhaus Dusseldorf, Düsseldorf, Germany
- Asian Institute of Gastroenterology, Somājigūda, Hyderabad, India
- Erasmus Medical Center, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No